CLINICAL TRIAL: NCT05904288
Title: Development of Digital Therapeutics Algorithms for Personalized Parkinson's Disease Treatment and Medication Plan Optimization
Brief Title: DTx Algorithms for Personalized Parkinson's Disease Treatment and Medication Plan Optimization
Status: Completed | Type: Observational
Sponsor: Newel Health SRL (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Other Study IDs: NWL-SOT-CS-001
Record Dates: First submitted 2023-05-08; First posted 2023-06-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Arm 1: The study group will receive noninvasive, in-depth clinical assessments similar in frequency to monitoring pertinent to normal clinical practice aimed at people with Parkinson's disease. In addition, within the mobile application provided as a gateway for data collection from the wearable sensors, subjects will also have the ability to access a library of video-recorded exercises, the effect of which on symptom modification, however, is not the subject of this investigation.
  Interventions: Device: Smartwatch Garmin Vivosmart [wearable sensor]; Device: Soturi™ [digital mobile app]; Other: Clinical Assessment

INTERVENTIONS:
Device: Smartwatch Garmin Vivosmart [wearable sensor] — Garmin Vivo Smart is a fitness tracker, which is aimed at collecting patient's motor activity and heart rate data from embedded Inertial Movement Unit (IMU) and Photoplethismograph (PPG) sensors.
Device: Soturi™ [digital mobile app] — Soturi software is a proprietary mobile application, for people with Parkinson's Disease (PD) designed to record symptoms, by means of self-report diary, set reminders for medication intake. Soturi™ Physical Exercise Program and Speech Exercise Program.
Other: Clinical Assessment — Outpatient repeated-measures clinical evaluations, which include assessment of motor symptoms through MDS-UPDRS and ecological motor tasks, to observe changes with respect to medication intake, and changes over a 6 month period time.

SUMMARY:
The study is aimed at developing Digital Therapeutics (DTx) algorithms for personalized PD treatment and medication plan optimization, based on Real World Data (RWD) collected from patients via digital mobile app and wearable sensors.

The study design is observational/noninterventional, prospective, single-arm, aimed at collecting data from wearable sensors for validation of symptom detection algorithms, through (1) a supervised in-clinic motor assessment, performed using validated clinical scales (Visit 3, Visit 4), and (2) an unsupervised, home-based, 6-month (Visit 3 to Visit 4) data collection from wearable devices (passive monitoring) for algorithm cross-validation using patient reported outcomes (PROMs) and remote clinical assessments. The devices used in the study will be a commercial smartwatch (Garmin Vivosmart 5) for inertial data collection and a digital application through which subjects will report PROMs via a digital symptom diary. Screening visits (Visit 1 and Visit 2) will be conducted prior to enrollment to verify eligibility criteria through clinical assessments, the subjects' symptom diary, and by assessing adherence to the use of the study tools provided (i.e., mobile application and smartwatch).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained.
2. Age > 18 years.
3. Male or female patients Meeting the MDS clinical diagnostic criteria for Parkinson's Disease (Postuma et al., 2015)
4. At least one motor symptoms OFF-period each day, excluding early morning akinesia.
5. On treatment with Levodopa
6. Stable Levodopa regimen for 4 weeks before Screening Visit;
7. Levodopa Equivalent Daily Dose (LEDD) > 400 mg, OR Levodopa Intake > 2 administration/day;
8. The subject is willing and able to attend study procedures and to use wearable and mobile devices.

Exclusion Criteria:

1. Secondary or atypical PD.
2. Cognitive problems which significantly impair his/her ability to give an IC and perform the study tasks.
3. Levodopa Equivalent Daily Dose (LEDD) > 800 mg, OR Levodopa intake > 8 administration/day;
4. Any condition that in the opinion of the investigator would interfere with the interpretation of the study results or constitute a health risk for the subject if he/she takes part in the study.
5. Concomitant participation to clinical trials with investigational medicinal products.
6. Failure to show, in opinion of the investigator, acceptable/appropriate use of wearable and mobile device (e.g. weekly average daily wearable wear time < 8 hours).

Having an advanced treatment (including Deep Brain Stimulation, Apomorphine, Duodopa), is not an exclusion criterion, as well as the subject decision or capability to attend the exercise and speech training programs within the mobile app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study targets individuals diagnosed with idiopathic PD which experience wearing-off phenomena.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Change in MDS-UPDRS Part III score from baseline to the 6-month follow-up visit, as measured during in-clinic visits. | Baseline to Week 26
  Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III includes 33 items to assess severity of motor symptoms, scoring per each item goes from 0= normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Total score ranges from 0 to 132.
Performance of the machine learning algorithm in predicting MDS-UPDRS Part III scores based on accelerometer data collected during in-clinic visits and home-based unsupervised data collected over 6 months. | Baseline to Week 26
  To develop and test machine learning model's performance outcome in predicting the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III motor symptoms scores.The specific outcome metrics and the respective units used to evaluate the models cannot be defined in advance, as they will depend on the nature of the data and the method of analysis as described by Giannakopoulou,et al. 2022 (Internet of Things Technologies and Machine Learning Methods for Parkinson's Disease Diagnosis, Monitoring and Management: A Systematic Review. Sensors, 22(5), 1799)
Change in patient-reported motor symptoms, as measured by an electronic symptoms diary, from baseline to the 6-month follow-up visit. | Baseline to Week 26
  "Change in Patient-Reported Motor Symptoms" focuses on assessing changes in motor symptoms reported by patients using an electronic symptoms diary, from baseline to the 6-month follow-up visit. Patients self-report their motor symptoms through the electronic diary, which allows them to record their symptoms and their severity, duration, and frequency.
Performance of the machine learning algorithm in predicting patient-reported symptom scores based on accelerometer data collected during in-clinic visits and home-based unsupervised data collected over 6 months | Baseline to Week 26
  To develop and test machine learning model's performance outcome in predicting patient-reported symptom scores. The specific outcome metrics and the respective units used to evaluate the models cannot be defined in advance, as they will depend on the nature of the data and the method of analysis as described by Giannakopoulou,et al. 2022 (Internet of Things Technologies and Machine Learning Methods for Parkinson's Disease Diagnosis, Monitoring and Management: A Systematic Review. Sensors, 22(5), 1799)

SECONDARY OUTCOMES:
Change in MDS-UPDRS Total Score and sub-scale total scores (Parts I-II-IV) | Baseline to Week 26
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a comprehensive assessment tool for Parkinson's disease. The MDS-UPDRS total scale, ranging from 0 to 199, measures the overall severity of motor and non-motor symptoms, with higher scores indicating worse outcomes. The subscales include Part I for non-motor aspects, Part II for motor aspects of daily living, Part III for motor examination, and Part IV for motor complications. Higher scores in all subscales suggest a worse outcome, reflecting the severity of symptoms in different domains.
Change in PDQ-39 Total Score | Baseline to Week 26
  The Parkinson's Disease Questionnaire-39 (PDQ-39) is a validated tool used to measure health-related quality of life in individuals with Parkinson's disease. With scores ranging from 0 to 100, higher scores on the PDQ-39 indicate a worse outcome. It assesses various domains, including mobility, activities of daily living, emotional well-being, stigma, social support, cognition, and communication. Higher scores reflect greater impairment and a lower quality of life, while lower scores indicate better overall well-being and functioning.
Change in Levodopa and Dopamine-Agonist Equivalent Daily Dosages (LEDD, DAEDD) | Baseline to Week 26
  "Change in Levodopa and Dopamine-Agonist Equivalent Daily Dosages (LEDD, DAEDD)" focuses on assessing the changes in the daily dosages of levodopa and dopamine agonists. Levodopa and dopamine agonists are common medications used in the treatment of Parkinson's disease. The dosages of these medications are calculated using standardized conversion factors to obtain Levodopa Equivalent Daily Dosage (LEDD) and Dopamine-Agonist Equivalent Daily Dosage (DAEDD), (expressed in mg/day). This outcome aims to measure any changes in the daily dosages of these medications over the course of the study or intervention.
Change in Levodopa Medication Plan: Medication Dose Strength | Baseline to Week 26
  "Change in Levodopa Medication Plan: Medication Dose Strength" focuses on assessing changes in the dose strength of levodopa medication per single intake event, measured in milligrams (mg).
Change in Levodopa Medication Plan: Units | Baseline to Week 26
  "Change in Levodopa Medication Plan: Units" focuses on assessing changes in the units of levodopa medication per single intake event. The units refer to the quantity of medication taken, which can be measured in whole pills, fractions of pills, or other specified units.
Change in Medication Levodopa Plan: Frequency of Intakes | Baseline to Week 26
  "Change in Medication Levodopa Plan: Frequency of Intakes" focuses on assessing changes in the frequency of intakes for a specified levodopa medication. The frequency refers to the total number of times the medication is taken in a day. Levodopa is a commonly prescribed medication for managing Parkinson's disease symptoms. This outcome aims to capture any modifications made to the frequency of intakes during the study or intervention period.
Change in Motor Symptoms Digital Biomarkers: duration | Baseline to Week 26
  "Change in Motor Symptoms Digital Biomarkers: duration" refers to the measure of time spent with specific motor symptoms. The duration is typically measured in minutes or seconds, representing the length of time an individual experiences the motor symptom being monitored. This outcome aims to capture any changes or fluctuations in the duration of motor symptoms over the course of the study or intervention.
Change in Motor Symptoms Digital Biomarkers: frequency | Baseline to Week 26
  "Change in Motor Symptoms Digital Biomarkers: frequency" focuses on measuring the frequency of motor symptoms experienced by individuals. The frequency is typically recorded as the number of occurrences within a specific time period, such as per hour or per day.
Change in Motor Symptoms Digital Biomarkers: severity | Baseline to Week 26
  "Change in Motor Symptoms Digital Biomarkers: severity" involves assessing the severity of motor symptoms using digital biomarkers on a scale ranging from 0 to 4.
Digital Biomarkers: Activity | Baseline to Week 26
  "Change in Digital Biomarker: Activity" measures the time spent on specific motor activities, such as walking, standing, active not moving, running, and climbing stairs, using digital biomarkers. The duration is measured in minutes and captures changes in activity time throughout the study or intervention.
Change in ePROMs: symptoms frequency | Baseline to Week 26
  "Change in ePROMs: Symptoms Frequency" uses the Soturi mobile app to collect electronic Patient-Reported Outcome Measures (ePROMs) regarding the frequency of symptoms. Participants report the frequency of specific symptoms they experience over time using the app.
Change in ePROMs: symptoms severity | Baseline to Week 26
  "Change in ePROMs: Symptoms Severity" utilizes the Soturi mobile app to collect electronic Patient-Reported Outcome Measures (ePROMs) regarding the severity of symptoms. Participants rate the severity of specific symptoms they experience on a scale ranging from 0 (absent) to 4 (severe) using the app.
Change in ePROMs, reported symptoms duration | Baseline to Week 26
  "Change in ePROMs: Symptoms Duration" involves using the symptom tracking function within the Soturi mobile app to collect electronic Patient-Reported Outcome Measures (ePROMs) regarding the duration of symptoms. Participants are asked to record the start time and end time of specific symptoms they experience using the app's symptom tracking feature.

OTHER OUTCOMES:
Usability of Soturi mobile app: System Usability Scale (SUS) | Baseline to Week 26
  "Usability of Soturi Mobile App: System Usability Scale (SUS)" assesses the usability of the Soturi mobile app using the System Usability Scale (SUS). The SUS is a validated questionnaire consisting of several statements related to app usability. Participants rate their agreement on a scale of 0 to 100, with higher scores indicating better usability. This outcome provides insights into the user-friendliness and effectiveness of the Soturi app. Higher scores on the SUS indicate a better outcome, suggesting that the app is more intuitive, easy to use, and meets user expectations. It helps evaluate and enhance the app's usability, resulting in improved user experiences and satisfaction
Usability of Soturi Mobile App: Session Duration | Baseline to Week 26
  "Usability of Soturi Mobile App: Session Duration" focuses on assessing the usability of the Soturi mobile app by analyzing session durations. Session duration refers to the length of time that users spend actively engaging with the app during a single session. By examining session durations, study will obtain insights into how long users typically interact with the app, indicating the level of engagement and usability. Longer session durations suggest that users find the app engaging and easy to navigate, indicating a positive usability outcome.
Usability of Soturi Mobile App: Frequency of App Interactions" | Baseline to Week 26
  "Usability of Soturi Mobile App: Frequency of App Interactions" assesses the usability of the Soturi mobile app by analyzing the frequency of user interactions. This outcome involves measuring how often users interact with different features and functions within the app. By analyzing the frequency of app interactions, study will determine the level of user engagement and the ease of navigating various app functionalities. A higher frequency of app interactions suggests that users find the app intuitive, engaging, and user-friendly, indicating a positive usability outcome.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Universitaria San Giovanni di Dio e Ruggi d'Aragona, Salerno, Salerno
  - IRCCS San Raffaele, Roma
  - IRCCS Fondazione Santa Lucia, Roma

IPD SHARING:
Plan to Share IPD: No